CLINICAL TRIAL: NCT02642315
Title: To Examine the Effect of Horizant (Gabapentin Enacarbil) in Primary Restless Legs Syndrome (RLS) Patients Who Are on Dopaminergic Agents and Exhibiting Augmentation
Brief Title: The Effect of Horizant (Gabapentin Enacarbil) on Augmentation
Acronym: XP-IIT-0034
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Pradeep Sahota, Professor & Chairman, Dept. of Neurology, University of Missouri-Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2002392
Record Dates: First submitted 2015-11-13; First posted 2015-12-30 (Estimated); Results first posted 2022-02-24 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Restless Legs Syndrome
MeSH Terms: conditions — Restless Legs Syndrome | interventions — Gabapentin; 1-(((alpha-isobutanoyloxyethoxy)carbonyl)aminomethyl)-1-cyclohexaneacetic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- open-label (Other): open-label single arm study
  Horizant, 600 mg oral once daily at 5 pm for 360 days.
  Interventions: Drug: Horizant

INTERVENTIONS:
Drug: Horizant — Phase1: During phase 1 therapy, Horizant will be added on as an adjunct to all subjects taking part in the study along with stable dose of their current dopaminergic (DA) agent and both medication will be continued for a total period of 90 days from day 0 to day 90. Subjects will be evaluated for three visits (days 0, 30 and 90) during Phase I.
  Phase 2: At the 90th day follow-up visit, with initiation of phase 2 therapy, all subjects will be tapered off (by 50% reduction in dose each week) of their current dopaminergic agents while maintaining the same dose of Horizant and will be on Horizant monotherapy. All subjects will be evaluated for additional three clinic visits (days 120, 180, 360).
  Other Names: Gabapentin enacarbil

SUMMARY:
Restless Legs Syndrome (RLS) is a common neurological disorder. Augmentation is the main complication during long-term DA treatment of RLS. This study aims to examine effect of Horizant (Gabapentin Enacarbil) on Augmentation in RLS patients.

DETAILED DESCRIPTION:
This is an Open label single arm study. The purpose of the study is to demonstrate the efficacy of Horizant in patients with RLS who exhibit augmentation while on Dopaminergic therapy. Adult patients (age 18-85 years) with diagnosis of primary RLS (diagnosed by study investigators) with augmentation on dopaminergic therapy will be screened for participation in the study. RLS diagnosis will be made by the study investigators using International RLS study group criteria. Patients with augmentation on dopaminergic therapy as defined by NIH 2007 with ASRS of 5 to 15 will be offered to participate in the study. Inclusion and exclusion criteria are listed below. The study will be performed after approval of the Institutional Review Board of the University of Missouri.

A total of 50 subjects will be entered into the study over a period of 1 year. Written consent will be obtained from all patients. After pre-participation evaluation for eligibility, subjects will be selected and enrolled in the study and followed for a total of 6 follow up visits (Days 0, 30, 90, 120, 180, 360). Subjects Enrollment period will last up to 12 months. The total duration of study will be 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients with diagnosis of RLS for more than one year.
2. Patients who are on DA therapy for 6 months or longer.
3. Patients who developed Augmentation (on stable dose of DA) lasting for 3 months or longer.
4. Augmentation severity rating scale of 5 to 15.
5. Both males and females
6. Age range = 18-85 year

Exclusion Criteria:

* Known Hypersensitivity to Horizant or Gabapentin products
* Peripheral neuropathy
* Radiculopathy
* Peripheral vascular disease
* Uremia [abnormal blood urea nitrogen (BUN) or Creatinine on Comprehensive Metabolic Panel (CMP)]
* Anemia
* Patients who are currently pregnant
* Patients who currently take opioids, lithium, anti-nausea medications (e.g. metoclopramide), dopaminergic antagonists (e.g. Haloperidol), 1st generation antihistamines (e.g. diphenhydramine, pseudoephedrine), anti-psychotic medications and iron therapy.
* Subjects with impaired decision making capability.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-01; Primary Completion 2019-05-06 (Actual); Study Completion 2019-05-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pradeep Sahota, MD, Principal Investigator — University of Missouri Health Care
Locations (1):
- University of Missouri Health Care, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Open-label: open-label single arm study
  Horizant, 600 mg oral once daily at 5 pm for 360 days.
  Horizant: Phase1: During phase 1 therapy, Horizant will be added on as an adjunct to all subjects taking part in the study along with stable dose of their current dopaminergic (DA) agent and both medication will be continued for a total period of 90 days from day 0 to day 90. Subjects will be evaluated for three visits (days 0, 30 and 90) during Phase I.
  Phase 2: At the 90th day follow-up visit, with initiation of phase 2 therapy, all subjects will be tapered off (by 50% reduction in dose each week) of their current dopaminergic agents while maintaining the same dose of Horizant and will be on Horizant monotherapy. All subjects will be evaluated for additional three clinic visits (days 120, 180, 360).
Period: Overall Study
Arm/Group | Open-label
Started | 10
Completed | 8
Not Completed | 2

BASELINE CHARACTERISTICS:
Population: Subjects:
  * Male and female patients
  * Ages 18 and 85
  * IRLS score
  * Augmentation Severity Rating Scale
Arm/Group | Open-label
Number analyzed (Participants) | 10
Age, Continuous [Median (Full Range); unit: years] | 54 [43 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
IRLS score [Median (Full Range); unit: units on a scale] — Higher International Restless Leg Syndrome - Rating Scale score means worse disease than lower score (Scale ranges from 1-40)
  units on a scale | 22.5 [13 to 28]
Augmentation Severity rating scale [Median (Full Range); unit: units on a scale] — Augmentation Severity Rating Scale:
  Higher number suggests worse disease than lower score (0-24)
  units on a scale | 7.5 [5 to 13]

OUTCOME MEASURES:

1. Primary Outcome: Change in Augmentation Severity From Day 0 to Day 90
Description: Augmentation severity rating scale; 0-24, 0 is better, 24 is worst
Time Frame: From Day 0 (Baseline) to Day 90
Population: 10 patients enrolled - 2 dropped out - 8 completed the study
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Open-label
Number analyzed (Participants) | 8
score on a scale
  Baseline | 6.5 [5 to 13]
  90 days | 0 [0 to 2]
Statistical Analysis 1: Comparison: Open-label; Test type: Other; p = 0.0131, Wilcoxon (Mann-Whitney); Median Difference (Net) = 36

2. Secondary Outcome: Change in Augmentation Severity Rating Scale Form Day 0 to Day 360 (270 Days After Discontinuation pf Dopaminergic Medication)
Description: Numeric Scale to assess degree of augmentation; Range 0-24; 0 is better, 24 is worst.
  We compared the Augmentation severity scale on day 0 to day 360 (which is 270 days after this decrease of dopaminergic medication)
Time Frame: Day 0 to day 360 (270 days after discontinuing dopaminergic medication)
Population: Only 8 subjects completed the study to its final point
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Open-label
Number analyzed (Participants) | 8
score on a scale
  Day 0 augmentation scale score | 6.5 [5 to 13]
  Day 360 Augmentation scale score | 0 [0 to 1]
Statistical Analysis 1: Comparison: Open-label; Test type: Other; p = 0.0131, Wilcoxon (Mann-Whitney); Median Difference (Net) = 36

ADVERSE EVENTS:
Time Frame: 1 year and 7 months
Description: Standard adverse event definition used
Arm/Group | Open-label
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 6/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-label (N=10)
Meralgia paraesthetica (Nervous system disorders) | 1 (1) — Meralgia paraesthetica
Hypertension (Cardiac disorders) | 1 (1)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Rheumatoid arthritis - exacerbation (Musculoskeletal and connective tissue disorders) | 1 (1)
Sleep apnea (Nervous system disorders) | 1 (1)
Calcification on right thyroid gland (Endocrine disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Limited (small numbers) open label study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-12-08): https://cdn.clinicaltrials.gov/large-docs/15/NCT02642315/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-08): https://cdn.clinicaltrials.gov/large-docs/15/NCT02642315/SAP_001.pdf